CLINICAL TRIAL: NCT01697579
Title: A Phase IIb, Partially-Blinded, Randomized, Active Comparator-Controlled Study to Evaluate the Pharmacokinetics/Pharmacodynamics, Safety, and Tolerability of Fosaprepitant in Pediatric Patients for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) Associated With Emetogenic Chemotherapy Sub-title: Open-Label Cohort to Further Evaluate the Pharmacokinetics/Pharmacodynamics, Safety, and Tolerability of Fosaprepitant in Pediatric Patients Birth to <12 Years Old
Brief Title: Study of the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Fosaprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Children (MK-0517-029)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0517-029; 2012-002340-24 (EudraCT Number); MK-0517-029 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant; Aprepitant; Injections; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Fosaprepitant 5 mg/kg-Cycle 1 (Experimental): Participants were administered intravenous (IV) fosaprepitant at the following weight-adjusted doses: participants 4 months to <12 years old were administered 5 mg/kg (not to exceed 150 mg); participants 1 to <4 months old were administered 2.5 mg/kg; participants 0 to <1 month old were administered 1.25 mg/kg. Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
  Interventions: Drug: Fosaprepitant; Drug: Ondansetron
- Fosaprepitant 3 mg/kg-Cycle 1 (Experimental): Participants 12 to 17 years old were administered 150 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 3 mg/kg (not to exceed 150 mg). Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
  Interventions: Drug: Fosaprepitant; Drug: Ondansetron
- Fosaprepitant 1.2 mg/kg-Cycle 1 (Experimental): Participants 12 to 17 years old were administered 60 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 1.2 mg/kg (not to exceed 60 mg). Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
  Interventions: Drug: Fosaprepitant; Drug: Ondansetron
- Fosaprepitant 0.4 mg/kg-Cycle 1 (Experimental): Participants 12 to 17 years old were administered 20 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 0.4 mg/kg (not to exceed 20 mg). Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
  Interventions: Drug: Fosaprepitant; Drug: Ondansetron
- Placebo Control-Cycle 1 (Placebo Comparator): Participants were administered IV normal saline at volume to match age and weight specific doses of fosaprepitant. Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
  Interventions: Drug: Fosaprepitant Placebo; Drug: Ondansetron
- Fosaprepitant 5 mg/kg-Cycles 2-6 (Experimental): For optional Cycles 2-6, participants from the 5 mg/kg fosaprepitant arm in Cycle 1 were administered fosaprepitant 5 mg/kg IV (or age-adjusted equivalent). For Cycle 2, fosaprepitant was administered IV plus ondansetron with or without dexamethasone. For Cycles 3-6, fosaprepitant was administered IV plus a 5- hydroxytryptamine 3 (5-HT3) antagonist with or without dexamethasone. Participants 1 year or less were required to receive ondansetron in all cycles as the 5-HT3 antagonist.
  Interventions: Drug: Fosaprepitant; Drug: 5-hydroxytryptamine 3 antagonist
- Fosaprepitant 3 mg/kg-Cycles 2-6 (Experimental): For optional Cycles 2-6, participants from Cycle 1 fosaprepitant arms (3, 1.2, or 0.4 mg/kg) or Cycle 1 control arm were administered fosaprepitant 3 mg/kg IV (or age-adjusted equivalent). For Cycle 2, fosaprepitant was administered IV plus ondansetron with or without dexamethasone. For Cycles 3-6, fosaprepitant was administered IV plus a 5-HT3 antagonist with or without dexamethasone.
  Interventions: Drug: Fosaprepitant; Drug: 5-hydroxytryptamine 3 antagonist

INTERVENTIONS:
Drug: Fosaprepitant — Administered intravenously (IV) as a single dose
  Other Names: Fosaprepitant dimeglumine; MK-0517; EMEND® for Injection
  Arms: Fosaprepitant 0.4 mg/kg-Cycle 1; Fosaprepitant 1.2 mg/kg-Cycle 1; Fosaprepitant 3 mg/kg-Cycle 1; Fosaprepitant 3 mg/kg-Cycles 2-6; Fosaprepitant 5 mg/kg-Cycle 1; Fosaprepitant 5 mg/kg-Cycles 2-6
Drug: Fosaprepitant Placebo — Administered IV as a single dose
  Arms: Placebo Control-Cycle 1
Drug: Ondansetron — Administered IV according to local labeling and/or local standard of care
  Other Names: Ondansetron hydrochloride; Zofran® Injection
  Arms: Fosaprepitant 0.4 mg/kg-Cycle 1; Fosaprepitant 1.2 mg/kg-Cycle 1; Fosaprepitant 3 mg/kg-Cycle 1; Fosaprepitant 5 mg/kg-Cycle 1; Placebo Control-Cycle 1
Drug: 5-hydroxytryptamine 3 antagonist — Administered IV according to local labeling and/or local standard of care
  Other Names: 5-HT3
  Arms: Fosaprepitant 3 mg/kg-Cycles 2-6; Fosaprepitant 5 mg/kg-Cycles 2-6

SUMMARY:
The purpose of this study was to determine the appropriate dosing regimen of fosaprepitant, when administered with ondansetron (with or without dexamethasone), for the prevention of CINV in children from birth to <17 years of age. Fosaprepitant is a prodrug to aprepitant. All participants who completed the randomized Cycle 1 could elect to receive open-label fosaprepitant during optional Cycles 2-6.

DETAILED DESCRIPTION:
Under Amendment 01, 0517-029 enrolled participants in the following age cohorts: 2-<6, 6-<12 and 12-17 years old. The study was randomized, partially-blinded, with parallel group assignment. Participants were randomized to one of three fosaprepitant doses or the control group. (Amendment 02 and Amendment 03 were country-specific amendments in Brazil that were required as per local regulations with no change in study design.) Under Amendment 04, the 12-17 year-old cohort was closed since that cohort fully enrolled. An additional fosaprepitant dose was added and all participants were allocated to this one treatment group. Amendment 04 was open-label and enrolled participants in the following age cohorts: 0-<2, 2-<6 and 6-<12 years old.

ELIGIBILITY:
Inclusion Criteria:

* Is 0 months (at least 37 weeks gestation) to <18 years of age
* Scheduled to receive chemotherapeutic agent(s) associated with moderate, high, or very high risk of emetogenicity for no more than 5 consecutive days for a documented malignancy, or a chemotherapy regimen not previously tolerated due to vomiting
* Expected to receive ondansetron as part of antiemetic regimen (Cycle 1); Expected to receive a 5-HT3 antagonist as part of antiemetic regimen (Cycles 2-6)
* If female and has begun menstruating, must have a negative pregnancy test prior to study participation and agree to remain abstinent or use a barrier form of contraception
* Predicted life expectancy of ≥3 months
* Pre-existing functioning central venous catheter
* Weight ≥3rd percentile for age and gender (and ≥3.0 kg)

Exclusion Criteria:

* Vomited in the 24 hours prior study drug administration (Cycle 1)
* Current user of any illicit drugs (including marijuana) or current evidence of alcohol abuse
* Scheduled to receive stem cell rescue therapy in conjunction with study related course(s) of emetogenic chemotherapy
* Received or will receive radiation therapy to the abdomen or pelvis in the week prior to study drug administration and/or during the course of the study
* Pregnant or breast feeding
* Allergic to fosaprepitant, aprepitant, ondansetron, or any other 5-HT3 antagonist
* Has a symptomatic central nervous system (CNS) tumor causing nausea and/or vomiting
* Has an active infection, congestive heart failure, slow heart rate, or other uncontrolled disease other than cancer
* Mentally incapacitated or has a significant emotional or psychiatric disorder
* Known history of QT prolongation or is taking any medication known to lead to QT prolongation
* Taking other excluded medications
* Participated in any previous study of aprepitant or fosaprepitant, or taken an investigational drug within 4 weeks prior to study participation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mora J, Valero M, DiCristina C, Jin M, Chain A, Bickham K. Pharmacokinetics/pharmacodynamics, safety, and tolerability of fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting in pediatric cancer patients. Pediatr Blood Cancer. 2019 Jun;66(6):e27690. doi: 10.1002/pbc.27690. Epub 2019 Mar 21. PMID 30900392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants scheduled to receive chemotherapeutic agent(s) associated with moderate, high, or very high risk of emetogenicity for no more than 5 consecutive days and were expected to receive ondansetron as part of their antiemetic regimen. Additional inclusion and exclusion criteria applied.
Pre-assignment Details: Participants (2 to <6, 6 to <12 and 12 to17 years-old) were enrolled in a randomized, partially-blinded study of 4 doses of fosaprepitant and a control in Cycle 1. Participants (0 to <2, 2 to <6 and 6 to <12 years-old) were invited to participate in optional Cycles 2-6 which was an open-label study of 2 doses of fosaprepitant.
Groups:
- Fosaprepitant 3 mg/Kg-Cycle 1: Participants 12 to 17 years old were administered 150 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 3 mg/kg (not to exceed 150 mg). Participants were also administered IV ondansetron 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 1.2 mg/Kg-Cycle 1: Participants 12 to 17 years old were administered 60 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 1.2 mg/kg (not to exceed 60 mg). Participants were also administered IV ondansetron 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 0.4 mg/Kg-Cycle 1: Participants 12 to 17 years old were administered 20 mg IV fosaprepitant. Participants 2 to <12 years old were administered a weight-adjusted dose of 0.4 mg/kg (not to exceed 20 mg). Participants were also administered IV ondansetron 0.15 mg/kg x 3 doses with or without dexamethasone.
Period: Base Study-Cycle 1
Arm/Group | Fosaprepitant 5 mg/Kg-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycle 1 | Fosaprepitant 1.2 mg/Kg-Cycle 1 | Fosaprepitant 0.4 mg/Kg-Cycle 1 | Placebo Control-Cycle 1 | Fosaprepitant 5 mg/Kg-Cycles 2-6 | Fosaprepitant 3 mg/Kg-Cycles 2-6
Started | 74 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6 arms.) | 43 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6 arms.) | 44 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6 arms.) | 41 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6 arms.) | 38 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6 arms.) | 0 (Enrollment in Cycles 2-6 was optional.) | 0 (Enrollment in Cycles 2-6 was optional.)
Completed | 72 | 42 | 43 | 40 | 35 | 0 | 0
Not Completed | 2 | 1 | 1 | 1 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Consent Withdrawn by Participant | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Optional Extension-Cycles 2-6
Arm/Group | Fosaprepitant 5 mg/Kg-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycle 1 | Fosaprepitant 1.2 mg/Kg-Cycle 1 | Fosaprepitant 0.4 mg/Kg-Cycle 1 | Placebo Control-Cycle 1 | Fosaprepitant 5 mg/Kg-Cycles 2-6 | Fosaprepitant 3 mg/Kg-Cycles 2-6
Started | 0 (47 participants from this arm in Cycle 1 entered optional Cycles 2-6 at 5 mg/kg) | 0 (33 participants from this arm in Cycle 1 entered optional Cycles 2-6 at 3 mg/kg) | 0 (25 participants from this arm in Cycle 1 entered optional Cycles 2-6 at 3 mg/kg) | 0 (27 participants from this arm in Cycle 1 entered optional Cycles 2-6 at 3 mg/kg) | 0 (21 participants from this arm in Cycle 1 entered optional Cycles 2-6 at 3 mg/kg) | 47 (Enrollment in Cycles 2-6 was optional.) | 106 (Enrollment in Cycles 2-6 was optional.)
Completed | 0 | 0 | 0 | 0 | 0 | 12 | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 35 | 69
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 1 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 7 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Excluded Medication | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Did Not Respond To Chemotherapy Regimen | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Completed Chemotherapy Regimen | 0 | 0 | 0 | 0 | 0 | 15 | 24
Not completed — Did Not Meet Cycle Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 4 | 11
Not completed — Consent Withdrawn by Participant | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Technical Problems | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Moved | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non-compliance With Protocol | 0 | 0 | 0 | 0 | 0 | 6 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant 5 mg/Kg-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycle 1 | Fosaprepitant 1.2 mg/Kg-Cycle 1 | Fosaprepitant 0.4 mg/Kg-Cycle 1 | Placebo Control-Cycle 1 | Total
Number analyzed (Participants) | 74 | 43 | 44 | 41 | 38 | 240
Age, Continuous [Mean (Standard Deviation); unit: Months] | 60.2 (42.3) | 123.8 (51.3) | 119.4 (52.7) | 119.2 (54.3) | 122.5 (54.0) | 102.4 (57.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 23 | 19 | 19 | 111
  Male | 42 | 25 | 21 | 22 | 19 | 129

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Aprepitant in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The Cmax for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: All participants 0 to <2 years of age that received one dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1: Participants were administered IV fosaprepitant at the following weight-adjusted doses: participants 4 months to <12 years old were administered 5 mg/kg (not to exceed 150 mg); participants 1 to <4 months old were administered 2.5 mg/kg; and participants 0 to <1 month old were administered 1.25 mg/kg. Participants were also administered IV ondansetron (0.15 mg/kg x 3 doses for children 6 months to 17 years of age or per local standard of care for children <6 months of age), with or without dexamethasone.
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 22
ng/mL | 3550 (1500)

2. Primary Outcome: Time to Maximum Concentration (Tmax) of Aprepitant in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The Tmax for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 22
hours | 2.01 (2.10)

3. Primary Outcome: Area Under the Concentration-time Curve of Aprepitant From Time 0 to Infinity (AUC 0-∞) in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The AUC 0-∞ for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 16
hr•ng/mL | 37200 (15800)

4. Primary Outcome: Area Under the Concentration-time Curve of Aprepitant From Time 0 to 24 Hours (AUC 0-24hr) in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The AUC 0-24hr for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 21
hr•ng/mL | 36800 (21800)

5. Primary Outcome: Apparent Terminal Half-life (t1/2) of Aprepitant in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The t1/2 for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 16
hours | 7.94 (2.86)

6. Primary Outcome: Concentration of Aprepitant After 24 Hours (C24hr) in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The C24hr for aprepitant was determined by measuring aprepitant levels in the time frame of 23 to 25 hours post-infusion.
Time Frame: Approximately 24 hours (from 23 to 25 hours) post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 21
ng/mL | 691 (852)

7. Primary Outcome: Concentration of Aprepitant After 48 Hours (C48hr) in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The C48hr for aprepitant was determined by measuring aprepitant levels in the time frame of 46 to 50 hours post-infusion. The C48hr was only planned to be measured in the 5 mg/mL dose for each age group.
Time Frame: Approximately 48 hours (from 46 to 50 hours) post-infusion
Population: All participants 0 to <2 years of age that received at least one 5 mg/mL dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 10
ng/mL | 352 (929)

8. Primary Outcome: Apparent Total Body Clearance (CL/F) of Aprepitant in Participants 0 to <2 Years of Age
Description: Fosaprepitant is a pro-drug that is rapidly converted to aprepitant. Because of this rapid conversion to aprepitant, fosaprepitant cannot be assessed directly. The pharmacokinetics for each fosaprepitant dose were determined by analyzing aprepitant in plasma. The CL/F for aprepitant was determined by measuring aprepitant levels at pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion.
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Fosaprepitant 5 mg/kg: 0 to <2 Years-Cycle 1
Number analyzed (Participants) | 16
mL/min | 24.2 (11.9)

9. Primary Outcome: Cmax of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 1
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: All participants 2 to <6 years of age that received one dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1: Participants were administered a weight-adjusted dose of 5 mg/kg fosaprepitant IV (not to exceed 150 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1: Participants were administered a weight-adjusted dose of 3 mg/kg fosaprepitant IV (not to exceed 150 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1: Participants were administered a weight-adjusted dose of 1.2 mg/kg of fosaprepitant IV (not to exceed 60 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1: Participants were administered a weight-adjusted dose of 0.4 mg/kg fosaprepitant IV (not to exceed 20 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 25 | 6 | 8 | 6
ng/mL | 4270 (2370) | 2320 (1540) | 2030 (1780) | 323 (103)

10. Primary Outcome: Tmax of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 2
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 25 | 6 | 8 | 6
hours | 1.90 (2.16) | 2.29 (2.14) | 1.36 (0.868) | 1.34 (0.771)

11. Primary Outcome: AUC 0-∞ of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 3
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 20 | 5 | 5 | 4
hr•ng/mL | 46400 (18600) | 15300 (11100) | 16000 (9680) | 2070 (992)

12. Primary Outcome: AUC 0-24hr of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 4
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 25 | 6 | 8 | 5
hr•ng/mL | 45000 (23800) | 21800 (22200) | 19700 (18500) | 1840 (742)

13. Primary Outcome: t1/2 of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 5
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 20 | 5 | 5 | 4
hours | 9.27 (4.17) | 6.55 (3.62) | 7.27 (3.47) | 6.18 (3.51)

14. Primary Outcome: C24hr of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 6
Time Frame: Approximately 24 hours (from 23 to 25 hours) post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 25 | 6 | 8 | 6
ng/mL | 1060 (1020) | 278 (398) | 332 (430) | 9.23 (14.8)

15. Primary Outcome: C48hr of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 7
Time Frame: Approximately 48 hours (from 46 to 50 hours) post-infusion
Population: All participants 2 to <6 years of age that received at least one 5 mg/mL dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 20 | 0 | 0 | 0
ng/mL | 232 (471) |  |  |

16. Primary Outcome: CL/F of Aprepitant in Participants 2 to <6 Years of Age
Description: as for outcome 8
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Fosaprepitant 5 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 2 to <6 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 2 to <6 Years-Cycle 1
Number analyzed (Participants) | 20 | 5 | 5 | 4
mL/min | 31.8 (13.8) | 66.2 (25.5) | 29.6 (22.1) | 48.5 (28.4)

17. Primary Outcome: Cmax of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 1
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: All participants 6 to <12 years of age that received one dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1: Participants were administered a weight-adjusted dose of 5 mg/kg fosaprepitant IV (not to exceed 150 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1: Participants were administered a weight-adjusted dose of 3 mg/kg fosaprepitant IV (not to exceed 150 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1: Participants were administered a weight-adjusted dose of 1.2 mg/kg of fosaprepitant IV (not to exceed 60 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1: Participants were administered a weight-adjusted dose of 0.4 mg/kg fosaprepitant IV (not to exceed 20 mg). Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 24 | 14 | 13 | 12
ng/mL | 4400 (1910) | 3550 (2460) | 1360 (903) | 507 (443)

18. Primary Outcome: Tmax of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 2
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 24 | 14 | 13 | 12
hours | 2.92 (5.09) | 1.99 (1.62) | 2.14 (1.96) | 1.68 (2.46)

19. Primary Outcome: AUC 0-∞ of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 3
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 13 | 8 | 9 | 8
hr•ng/mL | 55300 (11900) | 34300 (20300) | 10700 (5440) | 2860 (1120)

20. Primary Outcome: AUC 0-24hr of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 4
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 23 | 14 | 13 | 12
hr•ng/mL | 47400 (17300) | 29200 (14300) | 12000 (11000) | 4260 (5040)

21. Primary Outcome: t1/2 of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 5
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 13 | 8 | 9 | 8
hours | 9.77 (2.49) | 7.69 (2.09) | 8.23 (1.83) | 6.58 (2.36)

22. Primary Outcome: C24hr of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 6
Time Frame: Approximately 24 hours (from 23 to 25 hours) post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 24 | 14 | 13 | 12
ng/mL | 1210 (1000) | 589 (433) | 219 (379) | 70.4 (136)

23. Primary Outcome: C48hr of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 7
Time Frame: Approximately 48 hours (from 46 to 50 hours) post-infusion
Population: All participants 6 to <12 years of age that received at least one 5 mg/mL dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 11 | 0 | 0 | 0
ng/mL | 164 (124) |  |  |

24. Primary Outcome: CL/F of Aprepitant in Participants 6 to <12 Years of Age
Description: as for outcome 8
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Fosaprepitant 5 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 3 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 6 to <12 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 6 to <12 Years-Cycle 1
Number analyzed (Participants) | 13 | 8 | 9 | 8
mL/min | 42.1 (12.7) | 69.2 (66.4) | 78.8 (39.1) | 89.6 (40.9)

25. Primary Outcome: Cmax of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 1
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: All participants 12 to 17 years of age that received one dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1: Participants were administered 150 mg of fosaprepitant IV. Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1: Participants were administered 60 mg of fosaprepitant IV. Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
- Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1: Participants were administered 20 mg of fosaprepitant IV. Participants were also administered IV ondansetron at 0.15 mg/kg x 3 doses with or without dexamethasone.
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 12 | 12 | 13
ng/mL | 3500 (972) | 1180 (408) | 582 (437)

26. Primary Outcome: Tmax of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 2
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 12 | 12 | 13
hours | 0.546 (0.144) | 0.722 (0.608) | 0.736 (0.561)

27. Primary Outcome: AUC 0-∞ of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 3
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 3 | 8 | 9
hr•ng/mL | 33800 (7180) | 12300 (4660) | 3500 (1430)

28. Primary Outcome: AUC 0-24hr of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 4
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 12 | 12 | 13
hr•ng/mL | 30400 (8290) | 9700 (4200) | 4820 (7240)

29. Primary Outcome: t1/2 of Aprepitant in Participants 12 to 17 Years of Age Hours
Description: as for outcome 5
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 3 | 8 | 9
hours | 10.5 (1.00) | 7.92 (1.38) | 8.27 (1.20)

30. Primary Outcome: C24hr of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 6
Time Frame: Approximately 24 hours (from 23 to 25 hours) post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 12 | 12 | 13
ng/mL | 735 (310) | 142 (86.4) | 101 (247)

31. Primary Outcome: C48hr of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 7
Time Frame: Approximately 48 hours (from 46 to 50 hours) post-infusion
Population: All participants 12 to 17 years of age that received at least one 5 mg/mL dose of study therapy, did not have important deviations from the study protocol, and had data that contributed to the outcome being measured.
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 0 | 0 | 0

32. Primary Outcome: CL/F of Aprepitant in Participants 12 to 17 Years of Age
Description: as for outcome 8
Time Frame: Pre-infusion, immediately after infusion, and 2-4, 5-7, 8-10, 23-25, and 46-50 hours post-infusion
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Fosaprepitant 3 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 1.2 mg/kg: 12 to 17 Years-Cycle 1 | Fosaprepitant 0.4 mg/kg: 12 to 17 Years-Cycle 1
Number analyzed (Participants) | 3 | 8 | 9
mL/min | 76.2 (16.2) | 91.7 (32.5) | 105 (29.0)

33. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE) in Cycle 1
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol specified procedure, whether or not considered related to the medicinal product/protocol specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE.
Time Frame: Up to 14 days postdose in Cycle 1
Population: All randomized participants who received at least one dose of study treatment in Cycle 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Fosaprepitant 5 mg/Kg-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycle 1 | Fosaprepitant 1.2 mg/Kg-Cycle 1 | Fosaprepitant 0.4 mg/Kg-Cycle 1 | Placebo Control-Cycle 1
Number analyzed (Participants) | 74 | 42 | 43 | 40 | 35
Percentage of participants | 87.8 | 83.3 | 90.7 | 80.0 | 77.1

34. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE) in Cycles 2-6
Description: as for outcome 33
Time Frame: Up to 14 days postdose for each cycle (Cycles 2-6)
Population: All randomized participants who received at least one dose of study treatment in Cycles 2-6.
Measure: Number; unit: Percentage of participants
Arm/Group | Fosaprepitant 5 mg/Kg-Cycles 2-6 | Fosaprepitant 3 mg/Kg-Cycles 2-6
Number analyzed (Participants) | 44 | 80
Percentage of participants | 93.6 | 75.5

ADVERSE EVENTS:
Time Frame: Up to 14 days after the dose of study drug for Cycles 1-6 (approximately up to 84 days total)
Description: AEs were reported for the All Patients as Treated Population that included all randomized participants who received at least one dose of study treatment. All AEs (serious and non-serious) were reported in Cycle 1. In Cycles 2-6, only serious AEs and non-serious AEs that were either drug-related AEs or led to discontinuation were reported. The participants who completed Cycle 1 (base study) were invited to participate in optional Cycles 2-6; there were no new participants enrolled.
Arm/Group | Fosaprepitant 0.4 mg/Kg-Cycle 1 | Fosaprepitant 1.2 mg/Kg-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycle 1 | Fosaprepitant 5 mg/Kg-Cycle 1 | Placebo Control-Cycle 1 | Fosaprepitant 3 mg/Kg-Cycles 2-6 | Fosaprepitant 5 mg/Kg-Cycles 2-6
Serious Adverse Events (participants affected / at risk) | 11/40 | 14/43 | 12/42 | 24/74 | 12/35 | 46/106 | 24/47
Other Adverse Events (participants affected / at risk) | 27/40 | 33/43 | 32/42 | 60/74 | 24/35 | 69/106 | 31/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant 0.4 mg/Kg-Cycle 1 (N=40) | Fosaprepitant 1.2 mg/Kg-Cycle 1 (N=43) | Fosaprepitant 3 mg/Kg-Cycle 1 (N=42) | Fosaprepitant 5 mg/Kg-Cycle 1 (N=74) | Placebo Control-Cycle 1 (N=35) | Fosaprepitant 3 mg/Kg-Cycles 2-6 (N=106) | Fosaprepitant 5 mg/Kg-Cycles 2-6 (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 10 (10) | 7 (8) | 13 (13) | 4 (4) | 26 (47) | 18 (32)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (9) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (13) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopaenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorous decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetitie (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
air embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant 0.4 mg/Kg-Cycle 1 (N=40) | Fosaprepitant 1.2 mg/Kg-Cycle 1 (N=43) | Fosaprepitant 3 mg/Kg-Cycle 1 (N=42) | Fosaprepitant 5 mg/Kg-Cycle 1 (N=74) | Placebo Control-Cycle 1 (N=35) | Fosaprepitant 3 mg/Kg-Cycles 2-6 (N=106) | Fosaprepitant 5 mg/Kg-Cycles 2-6 (N=47)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 11 (12) | 12 (12) | 27 (28) | 10 (10) | 33 (54) | 14 (18)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 6 (6) | 5 (8) | 4 (4) | 10 (22) | 6 (16)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 10 (10) | 9 (10) | 18 (19) | 8 (8) | 14 (19) | 4 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 6 (7) | 11 (11) | 11 (11) | 9 (9) | 19 (44) | 10 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 6 (11) | 4 (6) | 6 (6) | 5 (5) | 4 (4) | 19 (30) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 9 (9) | 4 (4) | 9 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 6 (6) | 1 (1) | 10 (10) | 4 (5)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (3) | 4 (5) | 8 (21) | 2 (2) | 23 (40) | 6 (8)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 8 (8) | 3 (4)
Vomiting (Gastrointestinal disorders) | 9 (9) | 5 (5) | 7 (8) | 14 (20) | 3 (3) | 30 (69) | 12 (17)
Mucosal inflammation (General disorders) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 6 (9) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (4) | 5 (6) | 8 (8) | 3 (4) | 13 (19) | 4 (8)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 1 (2) | 6 (6) | 2 (3) | 15 (22) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 2 (4) | 8 (8) | 2 (2) | 13 (21) | 4 (5)
Neutrophil count decreased (Investigations) | 3 (3) | 5 (5) | 2 (3) | 11 (11) | 2 (2) | 15 (38) | 11 (17)
Platelet count decreased (Investigations) | 3 (3) | 7 (8) | 5 (5) | 16 (16) | 3 (3) | 15 (37) | 5 (8)
White blood cell count decreased (Investigations) | 5 (5) | 3 (5) | 2 (3) | 5 (5) | 3 (3) | 13 (23) | 5 (6)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 5 (8) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 3 (3) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 15 (25) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 9 (18) | 2 (3)
Headache (Nervous system disorders) | 3 (5) | 6 (9) | 4 (7) | 2 (2) | 2 (2) | 11 (15) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 6 (6) | 1 (1) | 12 (13) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 3 (5) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.